CLINICAL TRIAL: NCT06637644
Title: Impella RP Flex Registry
Brief Title: Impella RP Flex with Smart Assist
Status: Recruiting | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Impella RP Flex Study
Record Dates: First submitted 2024-09-18; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Right Ventricular (RV) Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients implanted with right-sided ventricular assist device
  Interventions: Device: Right-sided ventricular assist device

INTERVENTIONS:
Device: Right-sided ventricular assist device — Percutaneous device for right heart support

SUMMARY:
To capture observational data of the Abiomed Impella RP Flex in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received mechanical circulatory support (MCS) with an Impella RP Flex will be considered eligible for the registry.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes sites from the US
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objectives | 1 year post implant
  Survival at hospital discharge, with follow-ups at 30 days, 90 days, and 1-year post-discharge of Impella RP patients from real-world surveillance data.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pima Heart and Vascular, Tucson, Arizona
  - Baptist Health Heart Failure and Transplant Institute, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - University of Southern California (Keck USC), Los Angeles, California
  - Advent Health Orlando, Orlando, Florida
  - Tampa General, Tampa, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Metropolitan Heart and Vascular Institute, Coon Rapids, Minnesota
  - Providence St. Patrick Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health/Lenox Hill Hospital, New York, New York
  - Montefiore Medical Center - Moses, The Bronx, New York
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Research Institute (Legacy Emanuel Medical Center), Portland, Oregon
  - Oregon Health and Science System, Portland, Oregon
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Medical City Heart Hospital Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Memorial Herman Texas Medical Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - MultiCare Institute for Research Innovation, Puyallup, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Froedtert Hospital (Medical College of Wisconsin), Milwaukee, Wisconsin